CLINICAL TRIAL: NCT03320798
Title: Impact of Neurological Diseases on the Prognosis of Bullous Pemphigoid: A Retrospective Study of 178 Patients
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2016Ao004
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Bullous Pemphigoid
Keywords: Bullous pemphigoid; neurologic disorders
MeSH Terms: conditions — Pemphigoid, Bullous; Nervous System Diseases | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group "Bullous pemphigoid": Patients consulting at dermatology department of Reims Teaching Hospital for bullous pemphigoid between 1997 and 2011.
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record

SUMMARY:
Bullous pemphigoid affects mainly elderly patients. It is often associated with neurologic disorders, which represent a major risk factor of the disease

DETAILED DESCRIPTION:
The aim was to determine whether neurologic disorders, especially dementia, influences outcome and mortality of patients with bullous pemphigoid.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting bullous pemphigoid using the following criteria: clinical features typical of BP with presence of at least three out of four well-established criteria of Vaillant et al., subepidermal blister on skin biopsy and deposits of IgG and/or C3 in a linear pattern along the epidermal basement membrane zone by direct IF
* patients consulting at dermatology department of Reims Teaching Hospital (France) between 1997 and 2011

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting bullous pemphigoid and consulting at dermatology department of Reims Teaching Hospital (France) between 1997 and 2011.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
neurological disease | Day 0
  neurological disease are dementia (Alzheimers disease or other dementia), Parkinson's syndrome and stroke. Diagnosis of dementia was carried out in several ways: after examination by a neurologist or geriatrician, when the Mini Mental State was less than or equal to 17 or in the presence of a demonstrated and clinically evident dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France